CLINICAL TRIAL: NCT01904175
Title: Registry Study of T Cell Depleted Allogeneic Non-Myeloablative Stem Cell Transplant Recipients
Brief Title: Registry Study of T Cell Depleted Allo Non-Myeloablative Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00041936
Record Dates: First submitted 2012-12-05; First posted 2013-07-22 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Hodgkin's Disease; Non Hodgkin's Lymphoma; Myeloma; Leukemia; Myelodysplasia
Keywords: Stem cell transplantation, non-myeloablative
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell; Leukemia; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reduced Intensity Allogeneic Transplant: Subjects undergoing a reduced intensity allogeneic stem cell transplant

SUMMARY:
Allogeneic transplantation is used to treat many malignant and non-malignant diseases. The investigators and others have shown that less toxic preparative regimens (reduced intensity or 'mini' transplants) allow reliable allogeneic engraftment and durable remissions, significantly broadening the population of patients who may be offered this therapy to those who are older and more infirmed. The field is now focusing on the period post transplant for approaches to immune recovery leading to improved outcomes.

The primary objective of this registry is to catalogue data from patients who undergo standard of care reduced intensity allogeneic transplantation.

DETAILED DESCRIPTION:
Subjects will have toxicity monitored and reported per the Center for International Blood and Marrow Transplant Research (CIBMTR) program standard and as required by law for bone marrow transplant (BMT) reporting in the USA. Data will be collected from physical exam, laboratory studies, radiographs that are performed for clinical purposes. The tests and procedures are not in addition or in excess of our standards for allogeneic transplant outside of this registry. Data about donors will also be collected.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Subjects ≥ 18 years of age undergoing a reduced intensity allogeneic transplant

Exclusion Criteria:

* Subjects < 18 years of age
* Subjects not undergoing nonmyeloablative or ablative allogeneic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age undergoing a reduced intensity allogeneic stem cell transplant
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Catalogue Data | 1 year
  Catalogue data from subjects who undergo standard of care reduced intensity allogeneic transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States